CLINICAL TRIAL: NCT04178915
Title: Study of Leukocyte Immunophenotype and the Lipid Transport System as Predictive Biomarkers of Severe Bacterial Infections
Status: Enrolling by invitation | Type: Observational
Sponsor: The Republican Research and Practical Center for Epidemiology and Microbiology (Other)
Collaborators: Belarusian State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: RRPCEM_bacterial
Record Dates: First submitted 2019-11-24; First posted 2019-11-26 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Sepsis; Infective Endocarditis; Pneumonia, Bacterial
MeSH Terms: conditions — Sepsis; Endocarditis; Pneumonia, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Heparinized whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with severe bacterial infections
  Interventions: Diagnostic Test: Bood leukocyte subsets; Diagnostic Test: The cholesterol content of the cell membrane of T-cells and monocytes

INTERVENTIONS:
Diagnostic Test: Bood leukocyte subsets — Determination of blood leukocyte subpopulations, myeloid suppressor cells of various origins, type 2 congenital lymphoid cells, depleted T cells, CD45RA+ CD45RB+ CD62L-IRC, T-cell differentiation stages (naive - memory cells - effector - terminally differentiated effectors), B cells (CD5+ B1 cells, CD11c+ ABC, differentiation stages: immature - naive - isotype-unswitched memory cells - isotype-switched memory cells - plasmoblast)
Diagnostic Test: The cholesterol content of the cell membrane of T-cells and monocytes — The cholesterol content of the cell membrane of T-cells and monocytes with flow cytometry analysis

SUMMARY:
Current study evaluates the relationship between cell immunity and lipid transport systems in patients with severe bacterial infections (on the model of pneumonia, infective endocarditis, sepsis) in order to develop new methods for predicting the course and outcome of severe bacterial infections.

DETAILED DESCRIPTION:
* To study the state of the immune system in patients with severe bacterial infections (on the model of pneumonia, infective endocarditis, sepsis): spontaneous and stimulated production of reactive oxygen species by blood neutrophils; spontaneous necroptosis, apoptosis and pyroptosis of neutrophils; the content of blood leukocyte subpopulations.
* Assess the clinical, biochemical status, state of the lipid transport system of patients with severe bacterial infections (in the model of pneumonia, infective endocarditis, sepsis), including determination of the cholesterol content in the cell membrane of T-cells and monocytes.
* To develop a method for predicting an unfavorable course and an algorithm for the treatment (immunocorrection) of severe bacterial infections (on the model of pneumonia, infectious endocarditis, sepsis) based on the determination of the clinical and immunological status, indicators of the lipid transport system and dysmetabolic disorders, and propose a correction method for the treatment of these diseases, supplementing existing clinical protocols (preparations of immunoglobulins, lipids for parenteral nutrition, possibly PCSK9 inhibitors).

ELIGIBILITY:
Inclusion Criteria:

* community-acquired pneumonia, severe course (according to IDSA / ATs criteria) and / or sepsis with different localization of the primary focus (SOFA> 2);
* the patient's ability to comply with the instructions of the research doctor and follow the procedures required by the test protocol;
* informed consent.

Exclusion Criteria:

* acute and chronic heart failure;
* renal failure;
* acute and chronic liver failure;
* taking medications of the statin group during the last month before the study;
* diabetes in the stage of clinical and metabolic decompensation;
* acute and chronic leukemia, severe anemia;
* pregnancy or lactation;
* HIV infection;
* drug addiction;
* immunosuppressive therapy;
* malignant neoplasms over the past 5 years.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients with acute bacterial infections
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Elena Fomina, Dr, Principal Investigator — Head of the laboratory, RSPCEM
Locations (1):
- The Republican Research and Practical Center for Epidemiology and Microbiology, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: Undecided